CLINICAL TRIAL: NCT01520948
Title: Behavioral Therapy to Treat Urinary Symptoms in Parkinson Disease
Acronym: BETTUR PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Atlanta VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Camille Vaughan, MD, Staff Physician, Atlanta VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7892W
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Urinary Incontinence; Nocturia
Keywords: Parkinson disease; Incontinence
MeSH Terms: conditions — Urinary Incontinence; Nocturia; Parkinson Disease | interventions — Behavior Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise-based behavioral therapy (Experimental): Pelvic floor muscle exercise-based behavioral therapy
  Interventions: Behavioral: Exercise-based behavioral therapy
- Behavioral control (Placebo Comparator): Mirrored Star Drawing
  Interventions: Behavioral: Behavioral control

INTERVENTIONS:
Behavioral: Exercise-based behavioral therapy — Pelvic floor muscle exercise training, bladder training, fluid management, constipation management
  Arms: Exercise-based behavioral therapy
Behavioral: Behavioral control — Mirrored star drawing
  Arms: Behavioral control

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by motor symptoms of tremor, slowness of movement, and stiffness, leading to progressive disability and loss of independence. Lower urinary tract symptoms (LUTS), including urinary incontinence (UI), urgency, and/or nocturia, are common non-motor symptoms that further diminish the already compromised quality of life for adults living with PD. Behavioral interventions for UI - including pelvic floor muscle exercise (PFME) therapy - have proven efficacy in randomized controlled trials and are free of side effects. Exercise-based behavioral therapy for UI requires individuals to learn a motor skill (PFME) and implement an adaptive behavioral strategy that incorporates the PFME to suppress urinary urgency and prevent UI.

We will conduct a two-site, randomized controlled trial to assess the efficacy of PFME-based behavioral therapy to treat urinary symptoms in adults with PD. After stratification by UI severity, PD severity, and gender, a group of 60 subjects (30 in each group) will be randomized to receive behavioral therapy or a behavioral control over 8 weeks in order to achieve a sample size of 50 individuals (25 in each group) who complete the study. A 6-month follow-up is planned in the treatment group.

We hypothesize that:

1. PD participants who are randomized to the exercise-based behavioral therapy group (Group A) will report a significant reduction in weekly frequency of UI episodes compared to PD participants in the behavioral control group (Group B). The primary outcome, frequency of UI, will be measured using a seven-day bladder diary.
2. Compared to PD participants in Group B, the reduction in UI frequency in Group A will be clinically meaningful as measured by a corresponding improvement on questionnaires of satisfaction and quality of life as well as a decline in other urinary symptoms including urgency and nocturia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease determined by a board-certified neurologist with specialty training in movement disorders
* ≥ 4 weekly episodes of UI and at least one episode per week associated with feelings of urgency, where urgency is defined as the complaint of a sudden compelling desire to void which is difficult to defer
* Willingness to attend clinic visits
* Willingness to keep 7-day bladder diaries throughout the study period

Exclusion Criteria:

* Significant cognitive impairment, as indicated by a Montreal Cognitive Assessment (MoCA) score of < 18.
* Inability to produce an interpretable 7-day bladder diary at baseline
* Previous intensive PFME training
* Clinically significant depression as measured by a Geriatric Depression Scale-Short Form score ≥ 10 which could affect motivation to fully engage in the intervention
* Use of an indwelling urinary catheter
* Bladder outlet obstruction defined as having been prescribed in-and-out catheterization in the past 12 months, having a post-void residual urine volume by bladder ultrasound of ≥ 200 mL or a peak voiding flow rate of ≤ 4 mL/min on a void ≥ 125 mL in volume
* Severe uterine prolapse past the vaginal introitus
* Poorly controlled diabetes defined by a hemoglobin A1c (HgbA1c) of >8.0%
* Chronic renal failure and on hemodialysis
* Poorly controlled congestive heart failure or poorly controlled chronic obstructive pulmonary disease on physical exam
* Genitourinary cancer with ongoing surgical or external beam radiation treatment
* Any unstable health condition expected to result in hospitalization or death within in the next 3 months as determined by principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Bladder diary | 1 week

SECONDARY OUTCOMES:
Quality of Life Questionnaire | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: E. Camille Vaughan, MD, MS, Principal Investigator — Atlanta VAMC/Emory University
Locations (2):
- United States (2):
  - Birmingham VAMC, Birmingham, Alabama
  - Atlanta VA Medical Center, Decatur, Georgia